CLINICAL TRIAL: NCT05571605
Title: Cerebrovascular Dysregulation in Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas, Denton, TX (Other)
Responsible Party: Principal Investigator, Justin Sprick, Assistant Professor, University of North Texas, Denton, TX
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB # 22-305
Record Dates: First submitted 2022-09-30; First posted 2022-10-07 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Diseases
Keywords: exercise; brain blood flow
MeSH Terms: conditions — Renal Insufficiency, Chronic; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two conditions:1) aerobic exercise training on a stationary bicycle, or 2) stretching and balance training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (Experimental): Participants will exercise 3 times a week on a stationary bicycle. Exercise intensity will begin at low levels (50% of maximal heart rate reserve) and increase as tolerated to a maximum of 80% of maximal heart rate reserve. Exercise time will progress from an initial 20 minutes per session to a maximum of 45 minutes per session.
  Interventions: Behavioral: Exercise
- Stretching (Placebo Comparator): Participants will undergo progressive whole body stretching and balance exercises. This type of low intensity exercise is designed not to increase heart rate but rather to improve joint mobility and the ability to perform activities of daily living. This will serve as the control group to the exercise group. The control group will come in for stretching sessions 3 times per week for 20-45 minutes.
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Exercise — Participants randomized to this arm will exercise on a stationary bicycle.
  Arms: Exercise Training
Behavioral: Stretching — Participants randomized to this arm will perform stretching and balance exercise.
  Arms: Stretching

SUMMARY:
The purpose of this study is to test whether or not regular exercise training may improve brain blood flow regulation in patients with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Prior research has shown that CKD patients have an increased risk of stroke and that impairments in brain blood flow regulation predict stroke in other chronic disease states. This study will test whether exercise training can improve brain blood flow regulation via improved dynamic cerebral autoregulation and cerebrovascular carbon dioxide reactivity in CKD. Participants will undergo exercise training on a stationary bicycle, or stretching exercises, 3 times per week for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

• Individuals with chronic kidney disease stages III-IV.

Exclusion Criteria:

* Heart failure
* Chronic obstructive pulmonary disease
* Uncontrolled hypertension or hypotension
* Pregnancy or plans to become pregnant
* Inability to exercise on a stationary bicycle
* Current participation in exercise more than 20 minutes twice per week

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Texas, Denton, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exercise Training | Stretching
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training | Stretching | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 68 (6) | 66 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 0 | 4 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure-Middle Cerebral Artery Blood Velocity Very Low Frequency Phase (Radians)
Description: Mean arterial pressure was measured via finger photoplethysmography. Middle cerebral artery blood velocity was measured via transcranial Doppler ultrasound. A transfer function analysis was performed on the mean arterial pressure and middle cerebral artery blood velocity data to derive mean arterial pressure-middle cerebral artery blood velocity very low frequency phase (radians)
Time Frame: Mean arterial pressure-middle cerebral artery blood velocity transfer function phase (radians) will be compared at baseline (week 0) and after completing the 12-week intervention (week 13).
Measure: Mean (Standard Deviation); unit: Radians
Arm/Group | Exercise Training | Stretching
Number analyzed (Participants) | 5 | 6
Radians
  Baseline | 1.38 (0.45) | 1.12 (0.64)
  Post-Training | 1.40 (0.55) | 1.60 (0.40)
Statistical Analysis 1: Comparison: Exercise Training vs Stretching; Test type: Other; p = 0.05, ANOVA

2. Primary Outcome: Mean Arterial Pressure-Middle Cerebral Artery Blood Velocity Very Low Frequency Gain (cm/s/mmHg)
Description: Mean arterial pressure was measured via finger photoplethysmography. Middle cerebral artery blood velocity data was measured via transcranial Doppler ultrasound. A transfer function analysis was performed on the mean arterial pressure and middle cerebral artery blood velocity data to derive mean arterial pressure-middle cerebral artery blood velocity gain (cm/s/mmHg).
Time Frame: Mean arterial pressure-middle cerebral artery blood velocity transfer function gain (cm/s/mmHg) will be compared at baseline (week 0) and after completing the 12-week intervention (week 13).
Measure: Mean (Standard Deviation); unit: Cm/s/mmHg
Arm/Group | Exercise Training | Stretching
Number analyzed (Participants) | 5 | 6
Cm/s/mmHg
  Baseline | 0.65 (0.31) | 0.67 (0.19)
  Post-Training | 0.77 (0.20) | 0.63 (0.24)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Exercise Training | Stretching
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT05571605/Prot_SAP_000.pdf